CLINICAL TRIAL: NCT01484756
Title: Combined Vitamins and Minerals Decrease Incidence of Upper Respiratory Tract Infections in Older Persons
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Trisakti University (Other)
Responsible Party: Principal Investigator, Rina K Kusumaratna, Combined vitamins and minerals decrease incidence of upper respiratory tract infections in older persons, Trisakti University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FK-RKK-2819
Record Dates: First submitted 2011-11-15; First posted 2011-12-02 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Upper Respiratory Tract Infection
Keywords: respiratory infection; independent elderly; zinc; vitamins
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Zinc; Vitamins; Cold Temperature

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- calcium carbonate 500 mg (Placebo Comparator): Control group received one daily tablet of calcium carbonate 500 mg for 6 months
  Interventions: Dietary Supplement: Placebo
- daily multi micronutrient supplement (Experimental): Experimental group received one daily multi micro-nutrient supplement tablet for 6 months
  Interventions: Dietary Supplement: daily multi micronutrient supplement

INTERVENTIONS:
Dietary Supplement: daily multi micronutrient supplement — Multi micro-nutrient supplement tablet containing 40 mg elemental zinc (as gluconate, 120 mg ascorbic acid, 6 mg beta-carotene, 15 mg alpha-tocopherol (as d-alpha-tocopheryl acid succinate, 400 micrograms folic acid in experimental group given daily for six months
  Other Names: Zinc and vitamins for respiratory infection in older persons
  Arms: daily multi micronutrient supplement
Dietary Supplement: Placebo — calcium carbonate 500 mg
  Arms: calcium carbonate 500 mg

SUMMARY:
Nutrient deficiency and immune dysfunction in older persons result in high prevalence of acute respiratory infection,which can lead to impaired nutritional status. The study objective was to determine the effect of multi micro-nutrient supplementation on nutritional and upper respiratory infection among apparently healthy community-dwelling elderly. The main hypothesis was whether daily multi micro-nutrient supplementation could reduce the incidence and prevalence of upper respiratory infection among apparently healthy community-dwelling older persons. Inclusion criteria were apparently independent healthy male and female older persons aged 60 years and over, not taking multi micro-nutrient supplementation over the last month. The study design was a community-based double-blind controlled trial involving 296 community-dwelling older persons aged 60 and above, in the Mampang Prapatan district, South Jakarta. Participants were randomized to receive either 40 mg elemental zinc (as gluconate), 120 mg ascorbic acid, 6 mg B-carotene, 15 mg alpha tocopherol (as d-alpha-tocopheryl acid succinate) and 400 micrograms folic acid (intervention group) or 400 mg calcium carbonate (control group). Supplements were taken daily for six months, from August 2008 to March 2009. Nutritional and health status were measured before and after supplementation. Poisson regression analysis was used to evaluate the effects of daily multi micro-nutrient supplementation on the incidence and prevalence of upper respiratory infection.

DETAILED DESCRIPTION:
Poor nutritional status of older persons may predispose them to increased risk of upper respiratory tract infection, which however should be amenable to reduction by multi micro-nutrient supplementation. For becoming a successful healthy aging individual, the interrelationship between endogenous and exogenous factors must be positive and balanced. Introducing multi micro-nutrients through supplementation is an alternative which ensures a balanced micro-nutrient intake for enhancing the immune response and at the same time possibly enhancing the quality of life of the healthy free-living elderly individual.

The role of nutritional intervention strategies have been shown to be beneficial in the prevention of infectious disease among the older population in order to reduce the burden of diseases, and also could prevent micro-nutrient deficiency and enhance immune response of older persons.

The present study is related to primary prevention activities which aim to enhance the health status of the subjects, in particular to reduce the incidence and prevalence rate of infectious diseases, especially of upper respiratory tract infection. Supplementation is operationally achievable for implementation at the health center and could be set within the existing programs for older persons.

ELIGIBILITY:
Inclusion Criteria:

* women and men aged 60 years and above
* apparently healthy
* independent
* not taking supplementation during the last month

Exclusion Criteria:

* dementia or uncontrolled hypertension
* physically handicapped
* post cataract extraction

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
upper respiratory infection | 6 months
  This study measures number of new episodes of upper respiratory infection per total days of observation

SECONDARY OUTCOMES:
upper respiratory infection | 6 months
  This study measures number of days with upper respiratory infection per total days of observation

CONTACTS AND LOCATIONS:
Overall Officials: Rina K Kusumaratna, Dr, Principal Investigator — Faculty of Medicina, Trisakti University
Locations (1):
- Faculty of Medicine, University of Indonesia, Jakarta, Jakarta Special Capital Region, Indonesia

REFERENCES:
- [Background] Avenell A, Campbell MK, Cook JA, Hannaford PC, Kilonzo MM, McNeill G, Milne AC, Ramsay CR, Seymour DG, Stephen AI, Vale LD. Effect of multivitamin and multimineral supplements on morbidity from infections in older people (MAVIS trial): pragmatic, randomised, double blind, placebo controlled trial. BMJ. 2005 Aug 6;331(7512):324-9. doi: 10.1136/bmj.331.7512.324. PMID 16081445
- [Background] Barringer TA, Kirk JK, Santaniello AC, Foley KL, Michielutte R. Effect of a multivitamin and mineral supplement on infection and quality of life. A randomized, double-blind, placebo-controlled trial. Ann Intern Med. 2003 Mar 4;138(5):365-71. doi: 10.7326/0003-4819-138-5-200303040-00005. PMID 12614088
- See also: Click here for more information about this study — http://www.univmed.org